CLINICAL TRIAL: NCT00654082
Title: A Placebo-Controlled, Randomized, Two-Way Cross-Over, Double-Blind, Flexible Dose, Multicenter Study to Evaluate the Efficacy and Safety of Viagra in Male Patients With Traumatic Spinal Cord Injury and Erectile Dysfunction
Brief Title: A Study Evaluating the Efficacy and Safety of Sildenafil in Men With Traumatic Spinal Cord Injury and Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A1481103
Record Dates: First submitted 2008-03-31; First posted 2008-04-07 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Spinal Cord Injury; Erectile Dysfunction; Spinal Cord Trauma; Injuries, Spinal Cord; Impotence
MeSH Terms: conditions — Spinal Cord Injuries; Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: sildenafil
- Arm 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sildenafil — sildenafil 50 mg tablet by mouth 1 hour prior to anticipated sexual activity, but not more than once daily (QD) for 6 weeks; after 2 weeks on treatment, doses could be escalated to 100 mg or reduced to 25 mg
  Arms: Arm 1
Drug: placebo — placebo tablet by mouth 1 hour prior to anticipated sexual activity, but not more than once daily (QD) for 6 weeks
  Arms: Arm 2

SUMMARY:
To demonstrate the efficacy, safety and tolerability of sildenafil administered orally, as required, approximately 1 hour prior to sexual activity to men with erectile dysfunction (ED) associated with spinal cord injury (SCI), as well as its effects on the quality of life (QoL) of these patients.

ELIGIBILITY:
Inclusion Criteria:

-Patients were men with spinal cord injury and erectile dysfunction

Exclusion Criteria:

-N/A

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2002-09; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who indicated a preference for either treatment and who said that the treatment improved their erections | Weeks 6 and 14

SECONDARY OUTCOMES:
Responses to the International Index of Erectile Function (IIEF) | Weeks 0, 6, 8, and 14
Responses to the Global Efficacy Assessment (GEA) Question | Weeks 0, 6, 8, and 14
Responses to questions on the Quality of Life (QoL) Questionnaire | Weeks 0, 6, 8, and 14
Responses to Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Questions | Weeks 0, 6, 8, and 14
Intercourse success rate derived from patient event log | Weeks 0, 6, 8, and 14

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Turkey (Türkiye) (5):
  - Pfizer Investigational Site, Bahçelievler, Istanbul
  - Pfizer Investigational Site, Balçova, İzmir
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Bursa
  - Pfizer Investigational Site, Konya

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481103&StudyName=A%20Study%20Evaluating%20the%20Efficacy%20and%20Safety%20of%20Sildenafil%20in%20Men%20with%20Traumatic%20Spinal%20Cord%20Injury%20and%20Erectile%20Dysfunction.